CLINICAL TRIAL: NCT04877782
Title: Boosting a Neuromodulatory System Relevant to Alzheimer's Disease to Enhance Memory
Brief Title: Modulating the Locus Coeruleus Function
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: University of Liege (Other)
Responsible Party: Sponsor
Other Study IDs: NL77066.068.21
Record Dates: First submitted 2021-04-20; First posted 2021-05-07 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Healthy Aging
Keywords: Healthy aging; Transcutaneous vagus nerve stimulation; Magnetic resonance imaging; Locus coeruleus; Memory and attention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy older participants: Healthy older participants receiving both stimulation conditions (experimental and placebo) randomized across scanning sessions.
  Interventions: Device: Transcutaneous vagus verne stimulation

INTERVENTIONS:
Device: Transcutaneous vagus verne stimulation — Non-invasive and short electrical stimulation by placing the stimulating electrode at the cymba conchae of the left ear. The reference electrode is placed near the left cymba conchae. It provides a light tingling, massaging feeling in the ear.

SUMMARY:
The purpose of this study is to investigate the impact of transcutaneous vagus nerve stimulation (tVNS) on specific brain regions involved in memory and attention processes.

tVNS is a non-invasive and non-pharmacological technique known for targeting the locus coeruleus, a small subcortical nucleus in the brain thought to be involved in the earliest stages of Alzheimer's disease. This nucleus also plays a role in numerous cognitive functions, comprising memory and attention.

DETAILED DESCRIPTION:
This study is an observational MRI study with a pseudo-randomized single blind cross-over design. The population consists of 30 healthy human volunteers from 60 to 80 years old. These healthy older individuals will be recruited from the community.

After being informed about the study protocol and the potential risks, subjects will be given 1 week to consider their participation.

All participants giving written informed consent will be included in the study. The first session will consist in neuropsychological assessments and a task practice session in the dummy scanner in order to get familiar with the environment. Participants meeting the eligibility criteria will be included for the next sessions.

The second and third sessions are MRI scanning sessions including transcutaneous vagus nerve stimulation. Both the placebo and experimental stimulation conditions will be randomized in a single-blind manner across scanning sessions.

About 7 to 10 weeks after each scanning session and at least 4 days previous to the next MRI session, participant will be asked to fill in an online memory test for assessing potential outlasting effects of the stimulation technique.

ELIGIBILITY:
Inclusion Criteria:

* Average neuropsychological test results in accordance with normative data corrected for age, education and sex
* No substantial memory complaints according to the participant
* Body mass index < 28
* Non-smoking
* Right handedness
* Average/high level of education (minimum 12 years of education)

Exclusion Criteria:

* Psychoactive medication use
* Abuse of alcohol and drugs
* Cognitive impairment due to alcohol/drug or other substances abuse
* Recent trans-meridian travel (<2months)
* Night shift work (<1year)
* Diabetes if not stable
* Hypo-/hyper-tension, hypo-/hyper-thyroid if not stable
* Hypo-tension due to autonomic dysfunction
* Recent (<5years) or present psychiatric or neurological disorders (anxiety, major depression, schizophrenia, bipolar disorder, psychotic disorder -or treatment for it-, epilepsy, stroke, Alzheimer's disease, Parkinson's disease, multiple sclerosis, brain surgery, brain trauma, electroshock therapy, kidney dialysis, Ménière's disease, brain infections)
* Major vascular disorders (e.g. stroke)
* History of cardiovascular disorders (e.g., severe heart failure, recurrent vasovagal syncopal episodes)
* Major valvular disorders (e.g., prosthetic valve or hemodynamically relevant valvular disease, unilateral or bilateral vagotomy)
* Contraindications for scanning (e.g., brain surgery, cardiac pacemaker, metal implants, claustrophobia, body tattoos, reduced vision even after appropriate optical correction)
* Contraindications for pupil measurements and light exposure (e.g., Cataracts, Glaucoma, detached retina's, eye surgery involving the muscle, penetrating eye wounds, use of cholinesterase inhibitors, anticholinergic eye drop use, droopy eyelids preventing eye measurement).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy older individuals participating in the study will be recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Pupillometry - Scan session 1 | During the first MRI scanning session (55 minutes)
  Measure of pupil size variations during functional tasks. It can be used as a proxy for measuring arousal-related state transitions in brain activity and it allows for a reliable detection of the locus coeruleus activity.
Pupillometry - Scan session 2 | During the second MRI scanning session (55 minutes)
  Measure of pupil size variations during functional tasks. It can be used as a proxy for measuring arousal-related state transitions in brain activity and it allows for a reliable detection of the locus coeruleus activity.
Blood oxygen level dependent (BOLD) response - Scan session 1 | During the first MRI scanning session (55 minutes)
  This BOLD signal reflects brain activity during the functional tasks. The study focuses on the BOLD-signal in the locus coeruleus and task-relevant networks during the memory and the vigilance tasks.
Blood oxygen level dependent (BOLD) response - Scan session 2 | During the second MRI scanning session (55 minutes)
  This BOLD signal reflects brain activity during the functional tasks. The study focuses on the BOLD-signal in the locus coeruleus and task-relevant networks during the memory and the vigilance tasks.

SECONDARY OUTCOMES:
Performance on the online memory task - Post-session 1 | Performed from home, 7 to 10 days after the first MRI session and at least 4 days prior to the second session.
  Total accuracy on the face-name association task (from 0 to 100%); Mean reaction time on the face-name association task (from 0 to 4 seconds).
  The higher the total accuracy and the lower the mean reaction time, the better the outcome measure.
Performance on the online memory task - Post-session 2 | Performed from home, 7 to 10 days after the second MRI session.
  Total accuracy on the face-name association task (from 0 to 100%); Mean reaction time on the face-name association task (from 0 to 4 seconds).
  The higher the total accuracy and the lower the mean reaction time, the better the outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi IL Jacobs, Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD during the study are to be shared with the lab's members and according to the pre-defined agreements between Maastricht University and the University of Liège.
Supporting Information: Study Protocol
Time Frame: Previously mentioned IPD and additional supporting information will be shared from the end of the study ad will be available for a time period of 15 years.
Access Criteria: Data will be accessible only by lab members, through an access to the encrypted server where all data are stored.
  All kind of analyses might be performed on the available data.